CLINICAL TRIAL: NCT01948674
Title: Cognitive Training in Adolescents During Treatment for Substance Use Disorders
Brief Title: Cognitive Stimulation in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Matthew Johnson, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00080023; R21DA034942 (NIH)
Record Dates: First submitted 2013-09-17; First posted 2013-09-23 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- computerized tasks- adaptive (Experimental)
  Interventions: Behavioral: Computerized tasks
- computerized tasks - nonadaptive (Active Comparator)
  Interventions: Behavioral: Computerized tasks

INTERVENTIONS:
Behavioral: Computerized tasks — The study will compare the effects of different methods of computerized mental stimulation. The intervention involves 25 sessions involving computerized cognitive tasks.

SUMMARY:
The purpose of this study is to see if computer tasks that challenge the brain (cognitively stimulating tasks) can improve memory and other types of thinking in adolescents and young adults who are being treated for substance use problems. The study will compare the effects of different versions of the computer tasks.

ELIGIBILITY:
Inclusion Criteria:

* age 14-21
* Diagnosis of substance use disorder (SUD) by DSM-IV criteria with marijuana as primary substance of abuse
* eligible for intensive outpatient treatment

Exclusion Criteria:

* Untreated psychiatric disorder that might make participation hazardous
* Any condition associated with severe cognitive impairment

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
working memory (change from baseline) | expected within 2 weeks after intervention

SECONDARY OUTCOMES:
timeline follow back (change from baseline) | expected within 2 weeks after intervention
delay discounting (change from baseline) | expected within 2 weeks after intervention
Stroop (change from baseline) | expected within 2 weeks after intervention
reading comprehension (change from baseline) | expected within 2 weeks after intervention
emotion regulation (change from baseline) | expected within 2 weeks after intervention
Go-No Go (change from baseline) | expected within 2 weeks after intervention
Global Appraisal of Individual Needs (change from baseline) | expected within 2 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Johnson, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Mountain Manor Treatment Center, Baltimore, Maryland, United States